CLINICAL TRIAL: NCT04885439
Title: NextSteps: A Supportive Care Program For Advanced Cancer Patients and Their Caregivers
Brief Title: NextSteps Intervention for Advanced Cancer Patients and Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Hoda Badr, Dr., Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-39002
Record Dates: First submitted 2021-05-10; First posted 2021-05-13 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Lung Cancer; Gastrointestinal Cancer
MeSH Terms: conditions — Lung Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NextSteps Intervention (Experimental): Patients and caregivers will each receive their own tailored manual and six weekly 45-minute telephone calls that correspond to the manual, delivered by a Masters level trained interventionist.
  Interventions: Behavioral: NextSteps
- Usual Medical Care (No Intervention): UMC consists of standard oncologic care for the patient from the point of diagnosis of advanced cancer.

INTERVENTIONS:
Behavioral: NextSteps — Intervention sessions are delivered by a Masters level trained interventionist. During sessions, the interventionist will: conduct the weekly symptom screen, review content, answer questions, ensure skills mastery through homework review, and work with participants to develop action plans and identify/overcome barriers to self-care/caregiving. Patients and caregivers will receive individual calls from the interventionist for sessions 1, 2, and 3, and participate together for sessions 4, 5, and 6 via speakerphone.
  Arms: NextSteps Intervention

SUMMARY:
This study seeks to test the efficacy of a psychosocial intervention to empower advanced cancer patients and their caregivers and improve their quality of life (QOL). The program, called NextSTEPS, provides skills training in six domains that are central to patient and caregiver QOL: self-care, stress management, symptom management, effective communication, problem-solving, and social support.

DETAILED DESCRIPTION:
In this study, 200 advanced cancer patients who are within one month of treatment initiation (baseline) and their caregivers will complete baseline surveys and be randomized to NextSTEPS or a usual medical care (UMC) condition. In addition to UMC, patients and caregivers in the NextSTEPS condition will each receive an intervention manual and six weekly 45-minute telephone counseling sessions with a trained interventionist. Patients and caregivers in both the NextSTEPS and UMC conditions will complete follow-up surveys at 8 weeks (primary endpoint), and 4 and 6 months post-baseline (secondary endpoints).

The specific aims are to:

1. Determine the impact of NextSTEPS on patient physical and emotional QOL, palliative care utilization, and satisfaction with care relative to UMC. We hypothesize that at 8 weeks (2 months), and 4 and 6 months, patients in NextSTEPS will have less symptom burden, less emotional distress, greater palliative care utilization, and greater satisfaction with care relative to patients in UMC.
2. Determine the impact of NextSTEPS on caregiver self-care, physical and emotional QOL, and satisfaction with care. We hypothesize that at 8 weeks, and 4 and 6 months, caregivers in NextSTEPS will report more self-care, better physical QOL, less emotional distress, and greater satisfaction with care relative to caregivers in UMC.

Secondary/exploratory aims and hypotheses are to:

Examine the effects of the NextSTEPS intervention on Self Determination Theory (SDT) constructs. We hypothesize that NextSTEPS will enhance patient and caregiver competence, autonomy, and relatedness.

Test whether the SDT constructs of competence, autonomy and relatedness mediate the effects of NextSTEPS on patient/caregiver outcomes as hypothesized.

Explore whether sociodemographic (e.g., age, gender), medical (e.g., disease stage, comorbidities), and relationship factors (e.g., whether the caregiver is a spouse/partner or other family member) moderate the effects of NextSTEPS on patient/caregiver competence, autonomy, and relatedness.

NextSTEPS fills an important service gap by providing education, skills training, and support to advanced cancer patients and their caregivers shortly after diagnosis. Home-based telephone delivery will facilitate dissemination and outreach. By empowering families with the skills they need to coordinate care and meet the challenges of advanced cancer together, NextSTEPS holds great promise for improving patient and caregiver QOL, and the quality of palliative and supportive care in cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has stage 3A, 3B, or 4 NSLC or extensive stage SCLC and is within one month of treatment initiation OR patient has Stage 4 GI cancer and is within one month of treatment initiation
2. patient is spending more than 50% of time out of bed on a daily basis as measured by an ECOG Performance Status rating of level 0, 1, or 2
3. patient has stable brain metastases and no limitation on hepatic or renal function
4. patient has a spouse/partner other or close family member who he/she defines as the primary caregiver
5. patient and caregiver are age 18 years or older
6. patient and caregiver have the ability to read and understand English at a sixth grade level, as determined by ability to understand the consent form
7. patient and caregiver can provide informed consent

Exclusion Criteria:

1. patient or caregiver is deaf or has significant hearing impairment and thus cannot use the telephone
2. patient is currently enrolled in hospice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Patient and Caregiver Depression | 2 months
  Patient Reported Outcomes Measurement Information System Depression 6 item Short form
Patient and Caregiver Anxiety | 2 months
  Patient Reported Outcomes Measurement Information System Anxiety 6 item Short form

SECONDARY OUTCOMES:
Patient and Caregiver Satisfaction with Care | 2 months, 4 months, and 6 months
  20-item Family Satisfaction with Care (FAMCARE) scale
Patient Symptom Burden | 2 months, 4 months, and 6 months
  M D Anderson Symptom Inventory
Patient and Caregiver Depression | 4 and 6 months
  Patient Reported Outcomes Measurement Information System Depression 6 item Short form
Patient and Caregiver Anxiety | 4 and 6 months
  Patient Reported Outcomes Measurement Information System Anxiety 6 item Short form

CONTACTS AND LOCATIONS:
Overall Officials: Hoda Badr, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States